CLINICAL TRIAL: NCT05365503
Title: Dissemination Strategies and Implementation Outcomes of Adolescent Character Strength Interventions.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shamiri Institute (Other)
Collaborators: Africa Mental Health Research and Training Foundation (Unknown); Harvard University (Other); Kenyatta University (Other); WU Vienna University of Economics and Business (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Templeton 2 Phase 2
Record Dates: First submitted 2022-04-25; First posted 2022-05-09 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Mental Health Disorder
Keywords: Depression; Anxiety
MeSH Terms: conditions — Mental Disorders; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Shamiri Intervention (Experimental): The Shamiri intervention group will recieve a brief character strength intervention that will be delivered over the span of 4 weeks. There will be four sessions each lasting one hour each.
  Interventions: Other: Shamiri Intervention

INTERVENTIONS:
Other: Shamiri Intervention — The first two sessions focus on the concept of growth mindset, the third session focuses on gratitude, and the fourth and final session focuses on values. In session one, participants are guided through a Growth mindset intervention designed to convey the idea that people and their situations can change for the better. In session two, group leaders introduce a discussion and activities about effective strategies for growth. Then, the group leaders introduce a framework for problem solving. In session three, group leaders emphasize the importance of verbalizing and consciously thinking about Gratitude, as well as its benefits for well-being. In the final session, participants are introduced to the concept of values. Participants discuss stories of culturally pertinent role models, with an emphasis on the values these individuals display, and how their values guided their life decisions and led to success and happiness.

SUMMARY:
The present research study will involve investigating the efficacy of large-scale dissemination models of evidence-based character strength interventions in secondary schools in Kenya. This intervention, derived from a previously tested intervention named Shamiri, or thrive in Kiswahili, uses positive psychology and accessible life skills to build individual resilience and wellness. This will be a one-arm trial with participants recruited from 20 secondary schools in Nairobi, Kiambu and Makueni counties. The investigators estimate a sample size of 3000 youth, working on an intention to treat basis. All interested participants will be admitted to the program, with no exclusion criteria applied. The investigators will report on the efficacy of character strength interventions on wellbeing and mental health outcomes. Further, the investigators will also assess the scalability and acceptability of the program post intervention. Additionally, the investigators will examine moderator effects on the participants, baseline attributes of the participants, and potentially the effects of candidate mediators on intervention effects.

DETAILED DESCRIPTION:
This is a dissemination study whose objective is to explore the effectiveness, acceptability, and scalability of the Shamiri intervention when implemented in a large-scale naturalistic dissemination study in Kenyan secondary schools. Specifically, this study has two broad goals: 1) to test the effectiveness of Shamiri on mental health and psychosocial outcomes when delivered naturalistically on a large scale through either a centralized and de-centralized (train the trainers) administration, and 2) to examine and measure outcomes of these large-scale dissemination models.

For goal 1, participants will receive Shamiri directly through the Shamiri team or through an implementation partner. The investigators will measure mental health and psychosocial outcomes to determine if these outcomes compare to those reported in prior RCTs of Shamiri. The investigators hypothesize that participants receiving Shamiri will experience similar improvements in mental health and psychosocial outcomes as reported in previous RCTs. The investigators don't have a priori hypothesis on whether the mode through which the participants receive the intervention will affect intervention outcomes.

To achieve goal 2, investigators measure the following implementation related outcomes: intervention fidelity, cost, sustainment, acceptability, penetration, and cost-effectiveness. The investigators hypothesize that the Shamiri intervention will achieve high ratings in all intervention outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be high school students in one of the selected schools.
* Participants must be between the ages of 12 to 21.

Exclusion Criteria:

* There will be no other exclusion criteria.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3000 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Change in anxiety symptoms from baseline to 1-month follow up | Baseline, 2-week mid-point, 4-week end-point, and 1-month follow-up
  Self-reported anxiety symptoms, measured by the Generalized Anxiety Disorder Screener
Change in depression symptoms from baseline to 1-month follow up | Baseline, 2-week mid-point, 4-week end-point, and 1-month follow-up
  Self-reported depression symptoms as measured by the Patient Health Questionnaire - 8
Change in perceived social support from baseline to 1-month follow up | Baseline, 2-week mid-point, 4-week end-point, and 1-month follow-up
  Self-reported sense of social support, measured by the Multidimensional Scale of Perceived Social Support, with a score range of 0-7, with higher scores indicating greater perception of social support
Change in self-reported well-being from baseline to 1-month follow up | Baseline, 2-week mid-point, 4-week end-point, and 1-month follow-up
  Self-reported wellbeing, as measured by the Engagement, Perseverance, Optimism, Connectedness and Happiness Measure of Adolescent Well-Being, with a score range of 1-5, higher scores meaning better well-being
Change in academic performance from baseline to 1-month follow up | Baseline (academic term pre-intervention) and up to 1-month post intervention
  Academic performance, as measured by the average grade achieved from the school term before the intervention, the school term during which the intervention takes place, and the last term for which academic grades are available.

SECONDARY OUTCOMES:
Change in self-reported secondary control from baseline to 1-month follow up | Baseline, 2-week mid-point, 4-week end-point, and 1-month follow-up
  Self-reported participant sense of secondary control, or the ability to adjust oneself to hardships in such a way as to control their subjective emotional impact, measured by the 6-item short form of the Secondary Control Scale for Children (score range of 0-18, higher scores indicating greater perceived secondary control)
Change in sense of meaning and purpose in life from baseline to 1-month follow up | Baseline, 2-week mid-point, 4-week end-point, and 1-month follow-up
  Self-reported sense of purpose and meaning in life, as measured by the Purpose in Life Scale-12, with a score range of 20-140, higher scores indicating greater perceived meaning in life
Change in gratitude from baseline to 1-month follow up | Baseline, 2-week mid-point, 4-week end-point, and 1-month follow-up
  Self-reported gratitude, measured by a 6-item version of the Gratitude Questionnaire, with a score range of 6-48, with higher scores indicating higher gratitude
Change in perceived control from baseline to 1-month follow up | Baseline, 2-week mid-point, 4-week end-point, and 1-month follow-up
  Self-reported sense of control over oneself and one's life, measured by the Perceived Control Scale for Children, with a score range of 0-24, with a higher score indicating higher perception of control over one's life
Change in mental well-being from baseline to 1-month follow up | Baseline, 2-week mid-point, 4-week end-point, and 1-month follow-up
  Self-reported mental well-being of participants measured by the Short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS), with a score range of 7-35, higher scores indicating higher positive mental well-being

CONTACTS AND LOCATIONS:
Overall Officials: Tom L Osborn, Principal Investigator — Shamiri Institute
Locations (3):
- Kenya (3):
  - Shamiri Institute, Kiambu, Central Province
  - Africa Mental health Research and Training Foundation, Makueni, Eastern Province
  - Shamiri Institute, Nairobi

IPD SHARING:
Plan to Share IPD: Yes
The investigators intend to share fully de-identified data through publications and upon request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: T.B.D.
Access Criteria: T.B.D.

DOCUMENTS (1):
  • Informed Consent Form (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/03/NCT05365503/ICF_000.pdf